CLINICAL TRIAL: NCT05881044
Title: Psychiatric and Social Impacts of In Vitro Fertilization.
Brief Title: Psychiatric and Social Impacts of IVF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Hanna Abd elmalak bakhet, Principal Investigator, Assiut University
Other Study IDs: Impacts of IVF
Record Dates: First submitted 2023-03-24; First posted 2023-05-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: In Vitro Fertilization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychiatric interview — 1. Psychiatric interview which include personal identification, present history, past history and family history
  2. Complete physical and Neurological Examination.
  3. Mini Neuropsychiatric Interview scale. (MINI): to diagnosis psychiatric disorders
  4. Symptom checklist 90(SCL 90)
  5. Quality of life questionnaire.
  6. Hamilton Depression scale.
  7. Hamilton Anxiety scale.
  8. Socioeconomic scale (A.El.Gilany,A.El.Wehady,and M.EL.Wasify)

SUMMARY:
To asses psychiatric impacts of In vitro fertilization.

DETAILED DESCRIPTION:
Infertility and its treatment represent a global health area of increasing importance. Individuals experiencing infertility represent around 8-10% of couples worldwide.

The demand for assisted reproduction techniques such as in-vitro fertilization (IVF) has increased in developed countries over the past decades, and is predicted to increase further in those to come .

This could be further boosted by numbers in resource-limited settings of the developing world, where an estimated 180 million couples are experiencing infertility.

The efficacy of IVF among the assisted fertility options has led an increasing number of individuals to seek this specific treatment. More than a half million babies are now born each year from IVF, as a result of over two million estimated annual treatment cycles . Yet it is also a relatively invasive and disruptive process that can be both physically and psychologically demanding .

Infertility itself has been associated with a higher prevalence of depression and anxiety, lower quality of life, and lower self-esteem .

The IVF process-which includes injectable medication and multiple blood tests, clinic appointments and procedures, waiting periods and anticipation of outcomes at each phase-may lead to further psychological stress. This can be exacerbated by disturbances to an individual's work and routine and the financial pressure of this costly treatment , and may be worse after multiple failed cycles .

ELIGIBILITY:
Inclusion Criteria:

* Couples who perform or planning or failed to perform in vitro fertilization.
* Age from 18y To 40y .

Exclusion Criteria:

* Couples with any Psychiatric disorders prior to marriage.
* Couples with any physical or mental handcapes.
* refusal of couples to give consent to join the study.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: 1. Psychiatric interview which include personal identification, present history, past history and family history
  2. Complete physical and Neurological Examination.
  3. Mini Neuropsychiatric Interview scale. (MINI): to diagnosis psychiatric disorders
  4. Symptom checklist 90(SCL 90)
  5. Quality of life questionnaire.
  6. Hamilton Depression scale.
  7. Hamilton Anxiety scale.
  8. Socioeconomic scale (A.El.Gilany,A.El.Wehady,and M.EL.Wasify)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of depression in couples with IVF . | Baseline
  Measurement of psychiatric aspects in patients who perform or plan to perform in vitro fertilization by psychometric scales for measurement of depression such as The Hamilton Depression Rating Scale (HAM-D or HDRS) depression scale.
  * Scores below 7 generally represent the absence or remission of depression.
  * Scores between 7-17 represent mild depression
  * Scores between 18-24 represent moderate depression
  * Scores 25 and above represent severe depression

REFERENCES:
- [Background] Mascarenhas MN, Flaxman SR, Boerma T, Vanderpoel S, Stevens GA. National, regional, and global trends in infertility prevalence since 1990: a systematic analysis of 277 health surveys. PLoS Med. 2012;9(12):e1001356. doi: 10.1371/journal.pmed.1001356. Epub 2012 Dec 18. PMID 23271957
- [Background] Kocourkova J, Burcin B, Kucera T. Demographic relevancy of increased use of assisted reproduction in European countries. Reprod Health. 2014 May 26;11:37. doi: 10.1186/1742-4755-11-37. PMID 24885428